CLINICAL TRIAL: NCT01361360
Title: Permissive Hypercapnia and Brain Development in Premature Infants
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Thrasher
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- control
- hypercapnia

SUMMARY:
In the US, every year approximately 30,000 infants are born very prematurely, with birth weight less than 1000 grams. These infants usually require ventilators to help them breath normally during the first few weeks of life. Although the ventilator is lifesaving, it can also injure the very fragile lungs of these infants. Thus, a ventilation strategy, called permissive hypercapnia (high carbon dioxide), is widely used to prevent lung injury. Importantly, there is new research showing that high carbon dioxide may cause brain injury. In our proposed research, we will use magnetic resonance imaging methods to evaluate the brain in 40 very premature infants at term-equivalent age (Half of them had permissive hypercapnia ventilation, the other half did not) to see if permissive hypercapnia has adverse effect on brain development.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants with birth weight 401-1000 g

Exclusion Criteria:

* Those with complex congenital anomalies, central nervous system malformations, chromosomal abnormalities, or hydrops fetalis

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants with birth weight 401-1000 g (gestational age < 30 weeks)
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
MRI | 0

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States